CLINICAL TRIAL: NCT01801735
Title: A Multicenter, Open-Label, Safety Study of Meloxicam SoluMatrix™ Capsules in Subjects With Osteoarthritis of the Knee or Hip
Brief Title: Study of Meloxicam Capsules in Subjects With Osteoarthritis of the Knee or Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL3-12-03
Record Dates: First submitted 2013-02-21; First posted 2013-03-01 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meloxicam Test Capsules (Experimental): One Capsule QD
  Interventions: Drug: Meloxicam Test Capsules

INTERVENTIONS:
Drug: Meloxicam Test Capsules

SUMMARY:
The purpose of this study is to evaluate the safety of Meloxicam SoluMatrix Capsules for up to 52 weeks in subjects with pain due to osteoarthritis (OA) of the knee or hip

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 40 years of age
* If a participant in the previous MEL3-12-02 study, completed the study and did not discontinue for lack of efficacy or safety
* Has a diagnosis of OA of the hip or knee with ongoing knee and/or articular hip pain
* Chronic user of nonsteroidal anti-inflammatory drugs (NSAIDs) and/or acetaminophen for OA pain
* If female and of childbearing potential, is nonlactating and nonpregnant

Exclusion Criteria:

* History of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any NSAIDs, including meloxicam
* Requires continuous use of opioid or opioid combination products to control OA pain of the knee or hip
* Clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease
* Significant difficulties swallowing capsules or unable to tolerate oral medication
* Has received any investigational drug (except Meloxicam SoluMatrix Capsules), device, or therapy within 30 days before Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Carmichael, California
  - Pismo Beach, California
  - Milford, Connecticut
  - DeLand, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Ormond Beach, Florida
  - Ponte Vedra, Florida
  - Newton, Kansas
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Crestview Hills, Kentucky
  - Brockton, Massachusetts
  - Traverse City, Michigan
  - Troy, Michigan
  - Hazelwood, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hartsdale, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Duncansville, Pennsylvania
  - Anderson, South Carolina
  - Clinton, South Carolina
  - Austin, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Meloxicam 10 mg: Participants were administered Meloxicam 10 mg once daily for up to 52 weeks.
Period: Overall Study
Arm/Group | Meloxicam 10 mg
Started | 600
Completed | 390
Not Completed | 210
Not completed — Adverse Event | 79
Not completed — Lack of Efficacy | 28
Not completed — Withdrawal by Subject | 27
Not completed — Protocol Violation | 25
Not completed — Lost to Follow-up | 15
Not completed — Non-compliance with Trial Drug | 13
Not completed — Physician Decision | 3
Not completed — Death | 1
Not completed — Other, including site closure | 19

BASELINE CHARACTERISTICS:
Arm/Group | Meloxicam 10 mg
Number analyzed (Participants) | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358
  Male | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 567
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race; therefore, some subjects are counted multiple times.
  participants
    American Indian or Alaska Native | 2
    Asian | 6
    Black or African-American | 73
    Native Hawaiian or Other Pacific Islander | 1
    White | 520
Weight [Mean (Standard Deviation); unit: kg] | 88.50 (18.28)
Height [Mean (Standard Deviation); unit: cm] | 169.56 (10.17)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.65 (5.02)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Meloxicam 10 mg as Assessed by the Incidence of Adverse Events From Baseline to Week 52 or Early Termination
Description: The safety of Meloxicam 10 mg was assessed by the number of subjects with treatment-emergent adverse events (TEAEs), severe TEAEs, serious adverse events, treatment-related TEAEs, and adverse events (AEs) leading to discontinuation and subjects who died.
Time Frame: Baseline to Week 52/Early Termination
Measure: Number; unit: participants
Arm/Group | Meloxicam 10 mg
Number analyzed (Participants) | 600
participants
  Subjects with at least 1 TEAE | 406
  Subjects with at least 1 severe TEAE | 23
  Subjects with at least 1 serious adverse event | 35
  Subjects with at least 1 treatment-related TEAE | 127
  Subjects with AEs leading to discontinuation | 79
  Subjects who died | 2

ADVERSE EVENTS:
Arm/Group | Meloxicam 10 mg
Serious Adverse Events (participants affected / at risk) | 35/600
Other Adverse Events (participants affected / at risk) | 65/600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Meloxicam 10 mg (N=600)
Anemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Lobar pneumonia (Infections and infestations) | 1
Meningitis bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung squamous cell carcinoma, stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Hemorrhagic cerebral infarction (Nervous system disorders) | 1
Fourth nerve paralysis (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Medical device removal (Surgical and medical procedures) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Meloxicam 10 mg (N=600)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Urinary tract infection (Infections and infestations) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is required to submit any materials describing the results of the study at the site to sponsor for review not less than 30 days prior to publication and agrees to remove any of the Sponsor's confidential information. Sponsor also retains right to delay publication for an additional 60 day period to allow time for filing of patent applications.